CLINICAL TRIAL: NCT01149265
Title: Randomised Controlled Trial of an Existing Online Support Group for Depression and Anxiety
Brief Title: Online Support Groups for Depression and Anxiety
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University College, London (Other)
Responsible Party: Dr Chris Barker, University College London
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UCL1376/001
Record Dates: First submitted 2010-06-22; First posted 2010-06-23 (Estimated); Last update posted 2010-07-21 (Estimated); Status verified 2010-07

CONDITIONS: Depression; Anxiety
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Online support group (Experimental)
  Interventions: Behavioral: Online support group
- Expressive writing (Active Comparator)
  Interventions: Behavioral: Expressive writing

INTERVENTIONS:
Behavioral: Online support group — Expressive writing involves people writing about their thoughts and feelings, often upsetting ones, for a short period of time.
  Arms: Online support group
Behavioral: Expressive writing — Online support groups are internet forums where like-minded people give and receive both informational and emotional support.
  Arms: Expressive writing

SUMMARY:
The purpose of this study is to determine the effectiveness of online support groups for anxiety and depression.

DETAILED DESCRIPTION:
In recent years the number of online support groups for conditions like depression and anxiety has grown rapidly. Millions of people are thought to be using them around the world. This research aims to help find out whether the use of online support groups is beneficial and to learn more about what happens in these groups.

This research will compare online support groups with expressive writing. Expressive writing involves people writing about their thoughts and feelings, often upsetting ones, for a short period of time. In online support groups giving and receiving support from others can be helpful while expressive writing about emotional issues can be cathartic.

1,000 participants will be recruited online from the UK, USA and Canada and randomly assigned to either an existing online support group or to an expressive writing condition.

ELIGIBILITY:
Inclusion Criteria:

* Self-defined depression & anxiety
* Resident in the UK, US or Canada
* Access to the internet

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2010-05; Primary Completion 2011-02 (Estimated); Study Completion 2011-02 (Estimated)

PRIMARY OUTCOMES:
The Center for Epidemiological Studies Depression Scale | Zero, three and six months

SECONDARY OUTCOMES:
Satisfaction with Life Scale | Zero, three and six months
The Medical Outcomes Study Social Support Survey | Zero, three and six months
Generalised Anxiety Disorder Assessment | Zero, three and six months
The Illness perception questionnaire | Zero, three and six months

CONTACTS AND LOCATIONS:
Overall Officials: Chris Barker, Principal Investigator — University College, London
Locations (1):
- University College London, London, United Kingdom

REFERENCES:
- [Derived] Dean J, Potts HW, Barker C. Direction to an Internet Support Group Compared With Online Expressive Writing for People With Depression And Anxiety: A Randomized Trial. JMIR Ment Health. 2016 May 17;3(2):e12. doi: 10.2196/mental.5133. PMID 27189142